CLINICAL TRIAL: NCT05427799
Title: The Influence of Daily Honey Consumption on Insulin Resistance in Obese Women With Insulin Resistance
Brief Title: The Influence of Daily Honey Consumption on IR in Obese Women With IR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdul Hameed Shoman Foundation (Unknown)
Responsible Party: Principal Investigator, Shatha Hammad, Assistant Professor, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/137
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Honey; Gels

STUDY DESIGN:
Intervention Model Description: a parallel, single-blind, randomized trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey (Experimental): Treatment with honey will extend for four months and the actual treatment phases will be preceded by a 2-week run-in period, in which the participants will be asked to refrain from honey consumption.
  During the six months intervention, a daily dose of 0.5 g/kg body weight of honey will be consumed by each participant. Participants will be provided with Mixed flora honey that will be obtained from local producers. The daily dose of treatments will be divided into two doses to simulate a natural pattern of consumption.
  All participants will be required to limit the consumption of caffeinated beverages to two beverages a day during the study periods.
  A nutritionist will calculate the energy requirement and provide dietary instructions and a nutritionally adequate, hypocaloric, balanced sample diet plan with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein will be individualized for each participant monthly.
  Interventions: Dietary Supplement: Honey
- Other carbohydrate alternatives (Placebo Comparator): Treatment with simple sugar alternatives (other carbohydrates, such as jell-o) will extend for four months and the actual treatment phases will be preceded by a 2-week run-in period, in which the participants will be asked to refrain from honey consumption, and during the study periods.
  A daily dose of 0.5 g/kg body weight of jell-O will be consumed by each participant and will be divided into two doses to simulate a natural pattern of consumption. Jell-O was selected as a source of sucrose with negligible phenolic capacity, which will serve as a control.
  All participants will be required to limit the consumption of caffeinated beverages to two beverages a day during the study periods.
  A nutritionist will calculate the energy requirement and provide dietary instructions and a nutritionally adequate, hypocaloric, balanced sample diet plan with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein will be individualized for each participant monthly.
  Interventions: Dietary Supplement: Other carbohydrate alternatives such as jell-o

INTERVENTIONS:
Dietary Supplement: Honey — A mixed flora honey that will be obtained from local producers. and will be consumed by a daily dose of 0.5 g/kg body weight of honey by each participant and will be divided into two doses.
  Arms: Honey
Dietary Supplement: Other carbohydrate alternatives such as jell-o — A daily dose of 0.5 g/kg body weight of Jell-O will be consumed by each participant and will be divided into two doses. Jell-O was selected as a source of sucrose with negligible phenolic capacity.
  Arms: Other carbohydrate alternatives

SUMMARY:
The main objective of the study is to evaluate the effects of daily honey consumption on insulin resistance as a preventive measure against diabetes. in women with insulin resistance.

DETAILED DESCRIPTION:
The prevalence rates of insulin resistance (IR) and its health consequences are increasing worldwide. The reputation of honey as a healthy alternative for sugar is largely accepted. Honey contains several bioactive constituents; however, its effect on IR measures and glycemic control is yet to be assessed. We aim to evaluate the effect of daily consumption of honey on IR and inflammatory status measures in obese women with insulin resistance in a free-living controlled intervention study. Sixty obese adult females with insulin resistance will be recruited from the community of the University of Jordan and from patients at the Endocrine unit at the University of Jordan Hospital. Participants will be randomly assigned into one of two treatment groups, honey group or jell-O group. Participants will consume a daily dose of 0.5 mg per kg of body weight of the prescribed treatment for 6 months. The effects of daily consumption of honey on IR, serum concentration of several inflammatory biomarkers, and body fatness will be evaluated. The results of this study would reveal the antidiabetic effect of the bioactive compounds in honey in insulin-resistant obese women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 19-45 years
* Obese (BMI >= 30 kg/m^2)
* Premenopausal

Exclusion Criteria:

* Individual who use any drug or supplements known to affect lipid, glucose for at least the last three months.
* Individual who previous insulin treatment
* Smokers
* Individual who have diabetes, kidney, liver, or hormonal diseases
* Individual who have significant weight changes > 5% during the past 6 months
* Women who are postmenopausal

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Obese women with insulin resistance
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Dietary intake | Change from Baseline at 4 months
  Participants will provide a 3-day food record. Dietary data will be analyzed for energy, macro- and micro-nutrients composition using the food processor SQL version 10.3.0 program (ESHA Research, Salem, Oregon).
Dietary intake (A daily treatment consumption) | Every day of the treatment period (4 months)
  A daily treatment consumption checklist will be filled by each participant using the mobile App.
Anthropometric measurements (Height) | On the first day
  Standing height, without footwear, will be taken using stadiometer to the nearest 0.1 cm.
Anthropometric measurements (Weight) | Change from Baseline at 4 months
  Weight will be measured using a calibrated digital scale to the nearest 0.1 kg. All participants will be measured in light clothing and without any heavy articles or footwear.
Anthropometric measurements (Waist circumference) | Change from Baseline at 4 months
  The average waist circumference will be calculated from 2 consecutive measurements at the midway between the lowest rib and iliac crest.
Anthropometric measurements (A body composition assessment) | Change from Baseline at 4 months
  A body composition assessment will be performed using InBody120 analyzer (InBody, CO.). Participants will be asked to remove any metal items and heavy clothes before scanning, and will be scanned barefoot and wearing light clothes. Participant positioning will be conducted in accordance with the operator's manual.A trained operator will assess body composition according to the manufacturer's instructions.
Biochemical measurements (OGTT) | Change from Baseline at 4 months
  OGTT (75 g of glucose) will be executed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws. During OGTT venous blood samples will be obtained at 0, 30, 60, 90 and 120 min for the determination of glucose and insulin.
Biochemical measurements (OHTT) | Change from Baseline at 4 months
  OHTT (75 g of honey) will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws. During OHTT venous blood samples will be obtained at 0, 30, 60, 90 and 120 min for the determination of glucose and insulin.
Biochemical measurements (Glucose level) | Change from Baseline at 4 months
  Glucose level test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (Insulin level) | Change from Baseline at 4 months
  Insulin level test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (HbA1C) | Change from Baseline at 4 months
  HbA1C test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (Adiponectin) | Change from Baseline at 4 months
  Adiponectin test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (C-reactive protein) | Change from Baseline at 4 months
  C-reactive protein test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (Triglyceride) | Change from Baseline at 4 months
  Triglyceride test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (Total cholesterol) | Change from Baseline at 4 months
  Total cholesterol test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.
Biochemical measurements (High density lipoprotein- cholesterol (HDL-C)) | Change from Baseline at 4 months
  High density lipoprotein- cholesterol (HDL-C) test will be performed following an overnight fast and the participants will be instructed to abstain from consuming caffeinated beverages as well as from any type of exercise for 12 hours prior to blood draws.

OTHER OUTCOMES:
Dietary intake (3-day food record) | At the beginning of the study
  Participants will provide a 3-day food record. Dietary data will be analyzed for energy, macro- and micro-nutrients composition using the food processor SQL version 10.3.0 program (ESHA Research, Salem, Oregon).

CONTACTS AND LOCATIONS:
Overall Officials: Shatha S Hammad, PhD, Principal Investigator — The University of Jordan
Locations (2):
- Jordan (2):
  - Jordan University Hospital, Amman, Amman, Jordan
  - The University of Jordan, Amman, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal OP, Pachauri A, Yadav H, Urmila J, Goswamy HM, Chapperwal A, Bisen PS, Prasad GB. Subjects with impaired glucose tolerance exhibit a high degree of tolerance to honey. J Med Food. 2007 Sep;10(3):473-8. doi: 10.1089/jmf.2006.070. PMID 17887941
- [Result] Abbey EL, Rankin JW. Effect of ingesting a honey-sweetened beverage on soccer performance and exercise-induced cytokine response. Int J Sport Nutr Exerc Metab. 2009 Dec;19(6):659-72. doi: 10.1123/ijsnem.19.6.659. PMID 20175433
- [Result] Abdulrhman M, El Hefnawy M, Ali R, Abdel Hamid I, Abou El-Goud A, Refai D. Effects of honey, sucrose and glucose on blood glucose and C-peptide in patients with type 1 diabetes mellitus. Complement Ther Clin Pract. 2013 Feb;19(1):15-9. doi: 10.1016/j.ctcp.2012.08.002. Epub 2012 Oct 9. PMID 23337559
- [Result] Abu Rajab, A., Takruri, H., Mishal, A., & Alkurd, R. Glycemic and Insulinemic Response of Different Types of Jordanian Honey in Healthy and Type 2 Diabetic Volunteers. Pakistan Journal of Nutrition, 2017; 16(2), 61-68.
- [Result] Ajibola A., Physico-Chemical and Physiological Values of Honey and Its Importance as a Functional Food, International Journal of Food Sciences and Nutrition, 2015;2(6):1-9.
- [Result] Al-Ismail K., Herzallah, S. M., &Rustom, A. S. Antioxidant activities of some edible wild mediterranean plants. Italian Journal of Food Science, 2007; 19(3).
- [Result] Alvarez-Suarez J.M. , Tulipani S., Romandini S., Bertoli E., and Battino M., Contribution of honey in nutrition and human health: a review, Mediterranean Journal of Nutrition and Metabolism, 2010;3(1):15-23.
- [Result] Bermudez V, Salazar J, Martinez MS, Chavez-Castillo M, Olivar LC, Calvo MJ, Palmar J, Bautista J, Ramos E, Cabrera M, Pachano F, Rojas J. Prevalence and Associated Factors of Insulin Resistance in Adults from Maracaibo City, Venezuela. Adv Prev Med. 2016;2016:9405105. doi: 10.1155/2016/9405105. Epub 2016 Aug 4. PMID 27579182
- [Result] Farakla I, Koui E, Arditi J, Papageorgiou I, Bartzeliotou A, Papadopoulos GE, Mantzou A, Papathanasiou C, Dracopoulou M, Papastamataki M, Moutsatsou P, Papassotiriou I, Chrousos GP, Charmandari E. Effect of honey on glucose and insulin concentrations in obese girls. Eur J Clin Invest. 2019 Feb;49(2):e13042. doi: 10.1111/eci.13042. Epub 2018 Nov 16. PMID 30368796
- [Result] Ferreres F., García-Viguera C., Tomás-Lorente F., and Tomás-Barberán F.A., Hesperetin: a marker of the floral origin of citrus honey, Journal of the Science of Food and Agriculture, vol. 61, no. 1, pp. 121-123, 1993.
- [Result] Giugliano D, Ceriello A, Paolisso G. Oxidative stress and diabetic vascular complications. Diabetes Care. 1996 Mar;19(3):257-67. doi: 10.2337/diacare.19.3.257. PMID 8742574
- [Result] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Result] Kumar S., Safi S. Z., Qvist R., and Ismail I. S., Effect of agonists of adenosine receptors on inflammatory markers in human Muller cells, Current Science, 2014;106(4):582-586.
- [Result] Li N, Brun T, Cnop M, Cunha DA, Eizirik DL, Maechler P. Transient oxidative stress damages mitochondrial machinery inducing persistent beta-cell dysfunction. J Biol Chem. 2009 Aug 28;284(35):23602-12. doi: 10.1074/jbc.M109.024323. Epub 2009 Jun 22. PMID 19546218
- [Result] Molan PC. A brief review of honey as a clinical dressing. Prim Intention. 1998;6:148-158.
- [Result] Moniruzzaman M, Khalil MI, Sulaiman SA, Gan SH. Advances in the analytical methods for determining the antioxidant properties of honey: a review. Afr J Tradit Complement Altern Med. 2011 Oct 2;9(1):36-42. doi: 10.4314/ajtcam.v9i1.5. eCollection 2012. PMID 23983317
- [Result] de Rekeneire N, Peila R, Ding J, Colbert LH, Visser M, Shorr RI, Kritchevsky SB, Kuller LH, Strotmeyer ES, Schwartz AV, Vellas B, Harris TB. Diabetes, hyperglycemia, and inflammation in older individuals: the health, aging and body composition study. Diabetes Care. 2006 Aug;29(8):1902-8. doi: 10.2337/dc05-2327. PMID 16873800
- [Result] Nemoseck TM, Carmody EG, Furchner-Evanson A, Gleason M, Li A, Potter H, Rezende LM, Lane KJ, Kern M. Honey promotes lower weight gain, adiposity, and triglycerides than sucrose in rats. Nutr Res. 2011 Jan;31(1):55-60. doi: 10.1016/j.nutres.2010.11.002. PMID 21310307
- [Result] Oliveira LS, Santos DA, Barbosa-da-Silva S, Mandarim-de-Lacerda CA, Aguila MB. The inflammatory profile and liver damage of a sucrose-rich diet in mice. J Nutr Biochem. 2014 Feb;25(2):193-200. doi: 10.1016/j.jnutbio.2013.10.006. Epub 2013 Nov 15. PMID 24445044
- [Result] Pasupuleti VR, Sammugam L, Ramesh N, Gan SH. Honey, Propolis, and Royal Jelly: A Comprehensive Review of Their Biological Actions and Health Benefits. Oxid Med Cell Longev. 2017;2017:1259510. doi: 10.1155/2017/1259510. Epub 2017 Jul 26. PMID 28814983
- [Result] Qi Q, Bray GA, Smith SR, Hu FB, Sacks FM, Qi L. Insulin receptor substrate 1 gene variation modifies insulin resistance response to weight-loss diets in a 2-year randomized trial: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Circulation. 2011 Aug 2;124(5):563-71. doi: 10.1161/CIRCULATIONAHA.111.025767. Epub 2011 Jul 11. PMID 21747052
- [Result] Rao P.V., Krishnan K.T., Salleh N., and Gan S.H., Biological and therapeutic effects of honey produced by honey bees and stingless bees: a comparative review, RevistaBrasileira de Farmacognosia. 2016;26(5):657-664.
- [Result] Riccardi G, Giacco R, Rivellese AA. Dietary fat, insulin sensitivity and the metabolic syndrome. Clin Nutr. 2004 Aug;23(4):447-56. doi: 10.1016/j.clnu.2004.02.006. PMID 15297079
- [Result] Roncal-Jimenez CA, Lanaspa MA, Rivard CJ, Nakagawa T, Sanchez-Lozada LG, Jalal D, Andres-Hernando A, Tanabe K, Madero M, Li N, Cicerchi C, Mc Fann K, Sautin YY, Johnson RJ. Sucrose induces fatty liver and pancreatic inflammation in male breeder rats independent of excess energy intake. Metabolism. 2011 Sep;60(9):1259-70. doi: 10.1016/j.metabol.2011.01.008. Epub 2011 Apr 12. PMID 21489572
- [Result] Safi SZ, Qvist R, Yan GO, Ismail IS. Differential expression and role of hyperglycemia induced oxidative stress in epigenetic regulation of beta1, beta2 and beta3-adrenergic receptors in retinal endothelial cells. BMC Med Genomics. 2014 May 30;7:29. doi: 10.1186/1755-8794-7-29. PMID 24885710
- [Result] Samuel VT, Shulman GI. Mechanisms for insulin resistance: common threads and missing links. Cell. 2012 Mar 2;148(5):852-71. doi: 10.1016/j.cell.2012.02.017. PMID 22385956
- [Result] Sattar N., Perry C.G., and Petrie J. R. Type 2 diabetes as an inflammatory disorder, The British Journal of Diabetes and Vascular Disease, 2003;3(1):36-41.
- [Result] Tartibian B, Maleki BH. The effects of honey supplementation on seminal plasma cytokines, oxidative stress biomarkers, and antioxidants during 8 weeks of intensive cycling training. J Androl. 2012 May-Jun;33(3):449-61. doi: 10.2164/jandrol.110.012815. Epub 2011 Jun 2. PMID 21636735
- [Result] Al-Waili NS. Natural honey lowers plasma glucose, C-reactive protein, homocysteine, and blood lipids in healthy, diabetic, and hyperlipidemic subjects: comparison with dextrose and sucrose. J Med Food. 2004 Spring;7(1):100-7. doi: 10.1089/109662004322984789. PMID 15117561
- [Result] Yaghoobi N, Al-Waili N, Ghayour-Mobarhan M, Parizadeh SM, Abasalti Z, Yaghoobi Z, Yaghoobi F, Esmaeili H, Kazemi-Bajestani SM, Aghasizadeh R, Saloom KY, Ferns GA. Natural honey and cardiovascular risk factors; effects on blood glucose, cholesterol, triacylglycerole, CRP, and body weight compared with sucrose. ScientificWorldJournal. 2008 Apr 20;8:463-9. doi: 10.1100/tsw.2008.64. PMID 18454257
- See also: Type 2 diabetes as an inflammatory disorder — https://www.researchgate.net/profile/Dan-Ziegler-2/publication/7848046_Type_2_Diabetes_As_An_Inflammatory_Cardiovascular_Disorder/links/00b7d53c5247b6501b000000/Type-2-Diabetes-As-An-Inflammatory-Cardiovascular-Disorder.pdf
- See also: Prevalence and Associated Factors of Insulin Resistance in Adults from Maracaibo City, Venezuela — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4989131/